CLINICAL TRIAL: NCT02025478
Title: A Pilot Study of Enteral Donor Human Milk in Young Children Receiving Bone Marrow Transplantation
Brief Title: Human Breastmilk in Children Receiving a Bone Marrow Transplant
Acronym: MILK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Mothers' Milk Bank Northeast (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-2412
Record Dates: First submitted 2013-09-05; First posted 2014-01-01 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Bone Marrow Transplant- Autologous or Allogeneic
Keywords: children; bone marrow transplant; autologous; allogeneic; breastmilk; hematopoietic stem cell transplantation (HSCT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enteral Donor Breastmilk (Experimental): * Donor breast milk will be pasteurized prior to use.
  * Given orally or by nasogastric (NG) or nasojejunal (NJ) tube.
  * Feeding will be supervised and will be advanced as quickly as tolerated with a goal of providing 40-50% of nutritional needs from the donor milk.
  * It is recognized that the volume of enteral feeds will need to be adjusted per patient tolerance.
  Interventions: Dietary Supplement: Breastmilk

INTERVENTIONS:
Dietary Supplement: Breastmilk — * A registered dietician will supervise milk provision, and additional calories will be provided by addition of the supplement Prolacta. To make 28 kcal/oz milk, 40 ml of Prolacta will be mixed with 60 ml human milk to make a total volume of 100 ml.
  * If a nursing mother enrolls on the study, maternal and not donor milk will be given in the maximum volume possible, with Prolacta supplementation if clinically indicated and recommended by the registered dietician.

SUMMARY:
The investigators hypothesize that children receiving human milk will maintain a greater diversity of helpful bacteria in their gut and have lower levels of inflammatory proteins in the blood compared with children not receiving human milk.

DETAILED DESCRIPTION:
The investigators hypothesize that the gut microbiota during bone marrow transplant could be influenced by administration of enteral donor breast milk. This study will attempt to address this hypothesis, by feeding donor breast milk to young children undergoing transplant, and serially comparing the gut micobiota in children receiving human milk, with those receiving conventional feeding.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 5 years old receiving transplant (autologous or allogeneic)
* Parents must give informed consent

Exclusion Criteria:

- Failure to meet inclusion criteria

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Percentage of lactobacillales | 21 days after transplant
  Bar charts to indicate types and percentage of bacteria in stool samples - will quantify the bacterial diversity using the Shannon index and bacterial chaos using the Bray-Curtis time index.

SECONDARY OUTCOMES:
Levels of pro-inflammatory cytokines | Weekly during study course; up to approximately one year
  Mean fold increase above baseline for each cytokine will be calculated and compared to controls
Incidence of bacteremia | through day 14 post transplant
  Frequency of bacterial sepsis to be compared against controls
Incidence of graft versus host disease (GVHD) | through study course; approximately one year
  Frequency of GVHD will be compared to controls

CONTACTS AND LOCATIONS:
Overall Officials: Stella Davies, MBBS, PhD, MRCP, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States